CLINICAL TRIAL: NCT04176757
Title: A Phase 1 Open-Label, Multicenter Study to Evaluate Biomarkers for ZN-c5 in Subjects With Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Breast Cancer
Brief Title: A Study of ZN-c5 in Participants With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeno Alpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c5-002
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZN-c5 (Experimental)
  Interventions: Drug: ZN-c5

INTERVENTIONS:
Drug: ZN-c5 — ZN-c5 study drug to be administered orally daily

SUMMARY:
This is a Phase 1 open-label, multicenter study to evaluate biomarkers for ZN-c5 in subjects with breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated ICF
2. Age ≥ 18 years of age, either gender
3. Females must be postmenopausal as defined by at least one of the following:

   1. Age ≥ 60 years;
   2. Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and follicle stimulating hormone levels within the local laboratory's normal reference range for postmenopausal females;
   3. Documented bilateral oophorectomy
4. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the breast
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
6. Adequate organ function defined as follows:

   1. Hematologic: Platelets ≥ 100 × 109/L; Hemoglobin ≥ 9.0 g/dL; Absolute neutrophil count ≥ 1.5 × 109/L (without platelet transfusion or any hematopoietic growth factors within previous 7 days of the hematologic laboratory values obtained at the Screening Visit)
   2. Hepatic: Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT)

      ≤ 2.5 × upper limit of normal (ULN); Total or conjugated bilirubin ≤ 1.5 × ULN
   3. Renal: Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 60 mL/min

Exclusion Criteria:

1. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days of the first administration of study drug
2. Treatment with another investigational drug or other intervention within 28 days before the first administration of study drug
3. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral medication, including any unresolved nausea, vomiting, or diarrhea that is CTCAE v.5.0 Grade > 1
4. Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of study Day 1
5. Uncontrolled inter-current illness
6. History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the Investigator would pose a risk to subject safety or interfere with the study evaluations, procedures, or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Corroborate the single agent Recommended Phase 2 Dose | Throughout the study, an average of 15 months

SECONDARY OUTCOMES:
Dose-biomarker relationship | Throughout the study, an average of 15 months
  Percentage positive of Immunohistochemistry (IHC) staining Estrogen Receptor (ER) as compare to baseline
Dose-biomarker relationship | Throughout the study, an average of 15 months
  Percentage positive of IHC staining Progesterone Receptor (PR) as compare to baseline
Dose-biomarker relationship | Throughout the study, an average of 15 months
  Percentage positive of IHC staining Ki-67 as compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Ptaszynski, MD, Study Director — Zeno Alpha Inc.
Locations (10):
- United States (5):
  - Site 3, Tucson, Arizona
  - Site 2, New York, New York
  - Site 4, Nashville, Tennessee
  - Site 1, Houston, Texas
  - Site 5, Seattle, Washington
- Australia (4):
  - Site 11, Liverpool, New South Wales
  - Site 9, Sydney, New South Wales
  - Site 10, Cairns, Queensland
  - Site 8, Richmond, Victoria
- Site 7, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No